CLINICAL TRIAL: NCT01281553
Title: Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Assess the Efficacy and Safety of R051619 (Cisapride Oral Suspension 0.2 mg/kg q.i.d.) for the Treatment of Symptomatic Gastro-Oesophageal Reflux Disease (GORD) in Infants and Children
Brief Title: A Study of Cisapride in Patients With Symptomatic Gastro-Oesophageal Reflux Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Portfolio/CDT Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR003952; CIS-INT-27
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Cisapride (PREPULSID); Placebo; Gastroesophageal Reflux Disease (GERD); Gastro-oesophageal Reflux Disease (GORD)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Cisapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Cisapride 0.2 mg/kg suspension q.i.d.for 8 weeks.
  Interventions: Drug: Cisapride
- 002 (Placebo Comparator): Placebo Suspension identical in appearance to cisapride q.i.d. for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Suspension identical in appearance to cisapride q.i.d. for 8 weeks.
  Arms: 002
Drug: Cisapride — 0.2 mg/kg suspension q.i.d.for 8 weeks.
  Arms: 001

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of cisapride with placebo in infants and children with gastro-oesophageal reflux disease (GORD).

DETAILED DESCRIPTION:
This is a double-blind (neither patient nor study staff will know the identity of the assigned treatment) study evaluate the effectiveness and safety of cisapride in patients with gastro-oesophageal reflux disease (GORD) (also referred to as gastroesophageal reflux disease [GERD[) compared to a placebo (a identical in appearance to cisapride but does not contain active drug). Patients will receive placebo or cisapride suspension at 0.2 mg/kg (volumn determined by patient weight) four times per day (q.i.d.) (15 minutes before feeding 3 times a day and at bedtime) orally (by mouth) for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GORD based on protocol-specified characteristics
* Failed the 1st of 5 stepwise treatments for GORD recommended by the European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN)
* Caregiver able to complete the I-GERQ-R questionnaire

Exclusion Criteria:

* Protocol-specified respiratory conditions requiring previous or current treatment with oral or intravenous corticosteroids (prior and concurrent use of inhaled corticosteroids is acceptable)
* Cause of vomiting/regurgitation other than GORD
* Prior history of cisapride intake

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2003-09; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Caregiver's assessment of infant pediatric GORD symptoms | Up to 8 weeks (56 days)

SECONDARY OUTCOMES:
The number and type of adverse events reported | From time of first dose to the last dose (up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.